CLINICAL TRIAL: NCT03005301
Title: The CX-DZ-Ⅱ Intelligent Electroacupuncture Instrument for Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016XL007
Record Dates: First submitted 2016-12-24; First posted 2016-12-29 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Acupuncture; Neck Pain
Keywords: electroacupuncture instrument
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Selected acupoints will be stimulated by the new intelligent electro-acupuncture instrument.
  Interventions: Device: intelligent electroacupuncture instrument
- Control group (Active Comparator): Selected acupoints will be stimulated by the Hwato electroacupuncture instrument.
  Interventions: Device: Hwato electroacupuncture instrument

INTERVENTIONS:
Device: intelligent electroacupuncture instrument — Choice of major points: GB20, GB21, EX-B2, GV14. Choice of adjunct points based on syndrome differentiation.
  Trial instrument of this study is the CX-DZ-Ⅱ type intelligent electroacupuncture therapeutic instrument.Choice of acupuncture needle: one-off stainless acupuncture needle, which is 25~40mm in length and 0.30~0,38mm in diameter.Waveform: continuous-wave with frequency of 120~250 times per minute and current intensity within patients' tolerance.Treatment time: each treatment time is 30 minutes.
  Arms: Experimental group
Device: Hwato electroacupuncture instrument — Choice of major points: GB20, GB21, EX-B2, GV14. Choice of adjunct points based on syndrome differentiation.
  The Hwato electroacupuncture treatment instrument. Waveform: continuous-wave with frequency of 120~250 times per minute and current intensity within patients' tolerance.
  Treatment time: each treatment time is 30 minutes.
  Arms: Control group

SUMMARY:
The present study is a prospective, two-center, randomized, controlled, open-label, non-inferiority trial evaluating the efficacy and safety of a new intelligent electroacupuncture instrument in treating neck pain caused by cervical spondylosis.

DETAILED DESCRIPTION:
A total of 160 eligible patients will be included in this trial and randomly assigned to experimental group and control group in a 1:1 ratio. In experimental group, selected acupoints will be stimulated by the new intelligent electro-acupuncture instrument; while for control group, electroacupuncture treatment will be accomplished by a pre-existing electro-acupuncture instrument. The duration of treatment will be 2 weeks. The primary outcome is the change of visual analog scale score after one course of treatment. The secondary outcomes are visual analog scale score after each treatment, the responder rate, drug-usage rate of non-steroidal antipyretic analgesics, the occurrence rate of adverse events, defect rate of instrument, and excellent rate of instrument.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years old.
* Subject is diagnosed with CS of neck type or nerve-root type by clinical and medical imaging examination.
* A history of recurrent episodes of neck pain (one or more neck pain per month lasting for more than 3 months).
* Pain intensity is more than 3 points on a VAS upon recruitment.
* Subject or his guardian comprehend the aims of this trial, promise not to accept other relative treatments during the trial, and sign the informed consent.

Exclusion Criteria:

* Subject has acute neck trauma.
* Previous medical history of neck trauma treated by surgery, or neurological deficit, or congenital and developmental spinal disorders, or systemic bone diseases, or systemic joint diseases (e.g. joint slippage).
* Subject is diagnosed with carotid artery dissection.
* Subject is unable to express clearly self-feelings (e.g. subject with severe cerebrovascular accident sequelae).
* Subject has infection in acupuncture region.
* A history of acupuncture treatment for neck pain in the previous 1 week.
* Use of non-steroidal antipyretic analgesics in the previous 3 days.
* Subject has to use central analgesics or narcotic analgesics (e.g. Tramadol, Morphine, Dolantin) during the period of clinic trial.
* Use of various ointments or medicinal liquors with functions of promoting blood circulation and/or easing pain.
* Use of oral and intravenous medicines with functions of opening blood vessels and providing nutrition to nerve.
* Combinations of severe systematic diseases (e.g. a history of myocardial infarction, or severe hepatic and renal dysfunction, or acute infectious diseases, or malignant tumors, or severe mental disturbance diseases in previous 12 months).
* Intolerance of acupuncture and electro-acupuncture.
* Allergy to acupuncture.
* Female in pregnancy or lactation.
* Subject participate other clinic trials in previous 3 months.
* Subject is considered to be unsuited to this trial by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The change of VAS scores from baseline to the completion of treatment | 0-2 weeks

SECONDARY OUTCOMES:
VAS score after each treatment | 0-2weeks
Responder rate | 0-2weeks
Use of non-steroidal antipyretic analgesics | 0-2weeks
Adverse events | 0-2weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yulan Ren, Professor, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (2):
- China (2):
  - Affliated Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen ZH, Liang FR, Yang MX, Li DH, Zhang Y, Ren YL. Effect and Safety of CX-DZ-II Intelligent Electroacupuncture Therapeutic Instrument for Neck Pain Caused by Cervical Spondylos: Study Protocol for A Randomized Controlled Trial. Chin J Integr Med. 2020 May;26(5):375-381. doi: 10.1007/s11655-019-3038-2. Epub 2019 Aug 1. PMID 31372917